CLINICAL TRIAL: NCT02242942
Title: A Prospective, Open-Label, Multicenter Randomized Phase III Trial to Compare The Efficacy and Safety of A Combined Regimen of Obinutuzumab and Venetoclax Versus Obinutuzumab and Chlorambucil in Previously Untreated Patients With CLL and Coexisting Medical Conditions
Brief Title: Comparison of the Treatments of Obinutuzumab + Venetoclax Versus Obinutuzumab + Chlorambucil in Patients With Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: AbbVie (Industry); German CLL Study Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO25323; 2014-001810-24 (EudraCT Number); CLL14
Record Dates: First submitted 2014-09-16; First posted 2014-09-17 (Estimated); Results first posted 2019-10-01 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Lymphocytic Leukemia, Chronic
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Chlorambucil; venetoclax; obinutuzumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Safety Run-in Obinutuzumab + Venetoclax (Experimental): Subjects received obinutuzumab for 6 cycles and venetoclax for 12 cycles. Cycles comprised of 28 days.
  Interventions: Drug: Venetoclax; Drug: Obinutuzumab
- Obinutuzumab + Chlorambucil (Experimental): Participants will receive obinutuzumab for 6 cycles and chlorambucil for 12 cycles. Cycles will comprise 28 days.
  Interventions: Drug: Chlorambucil; Drug: Obinutuzumab
- Obinutuzumab + Venetoclax (Experimental): Participants will receive obinutuzumab for 6 cycles and venetoclax for 12 cycles. Cycles will comprise 28 days.
  Interventions: Drug: Venetoclax; Drug: Obinutuzumab

INTERVENTIONS:
Drug: Chlorambucil — Chlorambucil 0.5 milligrams per kilogram (mg/kg) orally at Day 1 and Day 15 at of each 28 day cycle for 12 cycles.
  Arms: Obinutuzumab + Chlorambucil
Drug: Venetoclax — Venetoclax, oral tablet: 20 mg daily during Cycle 1, Day 22-28; 50 mg daily during Cycle 2, Day 1-7; 100 mg daily during Cycle 2, Day 8-14; 200 mg daily during Cycle 2, Day 15-21; 400 mg daily during Cycle 2, Day 22-28 and on Day 1-28 for all subsequent cycles until the end of Cycle 12.
  Other Names: ABT-0199, GDC-0199
  Arms: Obinutuzumab + Venetoclax; Safety Run-in Obinutuzumab + Venetoclax
Drug: Obinutuzumab — Obinutuzumab, IV infusion: 100 mg or 1000 mg, depending on splitting rules, at Cycle 1, Day 1 (if 100 mg was received on Day 1, 900 mg will be administered on Cycle 1, Day 2); 1000 mg at Cycle 1, Day 8 and Day 15; 1000 mg at Day 1 for all subsequent cycles until the end of Cycle 6
  Other Names: GA-101; Gazyva

SUMMARY:
This open-label, multicenter, randomized Phase III study is designed to compare the efficacy and safety of a combined regimen of obinutuzumab and venetoclax versus obinutuzumab + chlorambucil in participants with chronic lymphocytic leukemia (CLL) and coexisting medical conditions. The time on study treatment was approximately one year and the follow-up period will be up to 9 years

ELIGIBILITY:
Inclusion Criteria:

* Documented previously untreated CLL according to the International Workshop on Chronic Lymphocytic Leukemia (IWCLL) criteria
* CLL requiring treatment according to IWCLL criteria
* Total Cumulative Illness Rating Scale (CIRS score) greater than (>) 6
* Adequate marrow function independent of growth factor or transfusion support within 2 weeks of screening as per protocol, unless cytopenia is due to marrow involvement of CLL
* Adequate liver function
* Life expectancy > 6 months
* Agreement to use highly effective contraceptive methods per protocol

Exclusion Criteria:

* Transformation of CLL to aggressive Non-Hodgkin's lymphoma (Richter's transformation or pro-lymphocytic leukemia)
* Known central nervous system involvement
* Participants with a history of confirmed progressive multifocal leukoencephalopathy (PML)
* An individual organ/ system impairment score of 4 as assessed by the CIRS definition limiting the ability to receive the treatment regimen of this trial with the exception of eyes, ears, nose, throat organ system
* Participants with uncontrolled autoimmune hemolytic anemia or immune thrombocytopenia
* Inadequate renal function
* History of prior malignancy, except for conditions as listed in the protocol if participants have recovered from the acute side effects incurred as a result of previous therapy
* Use of investigational agents or concurrent anti-cancer treatment within the last 4 weeks of registration
* Participants with active bacterial, viral, or fungal infection requiring systemic treatment within the last two months prior to registration
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies or known sensitivity or allergy to murine products
* Hypersensitivity to chlorambucil, obinutuzumab, or venetoclax or to any of the excipients
* Pregnant women and nursing mothers
* Positive test results for chronic hepatitis B virus (HBV) infection (defined as positive hepatitis B surface antigen [HBsAg] serology) or positive test result for hepatitis C (hepatitis C virus [HCV] antibody serology testing)
* Participants with known infection with human immunodeficiency virus (HIV) or human T-cell leukemia virus-1 (HTLV-1)
* Requires the use of warfarin, marcumar, or phenprocoumon
* Received agents known to be strong and moderate Cytochrome P450 3A inhibitors or inducers within 7 days prior to the first dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 445 (Actual)
Dates: Start 2014-12-31 (Actual); Primary Completion 2018-08-17 (Actual); Study Completion 2025-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (122):
- United States (8):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - City of Hope, Duarte, California
  - UC San Diego Health System, La Jolla, California
  - Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute, Atlanta, Georgia
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Henry Ford Hospital, Detroit, Michigan
  - Joe Arrington Cancer Center, Lubbock, Texas
- Hospital Italiano, Buenos Aires, Argentina
- Australia (9):
  - Liverpool Hospital, Liverpool BC, New South Wales
  - Tweed Hospital, Tweed Heads, New South Wales
  - The Townsville Hospital, Douglas, Queensland
  - Princess Alexandra Hospital Woolloongabba, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Ashford Cancer Centre Research, Ashford, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - The Northern Hospital, Epping, Victoria
  - Monash Medical Centre, Melbourne, Victoria
- Austria (3):
  - Tiroler Landeskrankenanstalten Ges.M.B.H., Innsbruck
  - Medizinische Universität Wien, Vienna
  - Hanusch-Krankenhaus, Vienna
- Brazil (4):
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
  - Instituto de Ensino e Pesquisa Sao Lucas - IEP, São Paulo, São Paulo
  - Hospital Sírio-Libanês, São Paulo, São Paulo
  - Hospital das Clinicas - FMUSP, São Paulo, São Paulo
- Bulgaria (5):
  - UMHAT Dr Georgi Stranski, Pleven
  - UMHAT " Sveti Georgi" Plovdiv - Clinic of Oncology and Hematology, Plovdiv
  - University Hospital Sv.Georgi Clnic of Hematology, Plovdiv
  - University Multiprofile Hospital For Active Treatment "Sveti Ivan Rilski" EAD, Sofia
  - MHAT Hristo Botev, Vratsa
- Canada (3):
  - Arthur J.E. Child Comprehensive Cancer Center, Calgary, Alberta
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Jewish General Hospital, Montreal, Quebec
- Croatia (2):
  - University Hospital Center Zagreb, Zagreb
  - University Hospital Merkur Clinic for Internal Medicine/ Hematology, Zagreb
- Denmark (4):
  - Herlev Hospital, Herlev
  - Rigshospitalet, København Ø
  - Sjaellands Universitetshospital, Roskilde, Roskilde
  - Sygehus Lillebælt, Vejle, Vejle
- Estonia (2):
  - North Estonia medical Centre, Tallinn
  - Tartu Uni Hospital, Tartu
- France (12):
  - Institut d'Hématologie de Basse Normandie, Caen
  - Hopital Henri Mondor, Créteil
  - CHU de Grenoble, Grenoble
  - Centre Jean Bernard, Le Mans
  - Centre Leon Berard, Lyon
  - Hôpital Saint Eloi, Montpellier
  - Hopital Hotel Dieu Et Hme, Nantes
  - Hopital Saint Louis, Paris
  - Hopital Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - CH de Toulon Hôpital Sainte Musse, Toulon
  - Institut Gustave Roussy - Hematologie, Villejuif
- Germany (24):
  - Uniklinik RWTH Aachen, Aachen
  - Charite - Campus Virchow-Klinikum, Berlin
  - Charite - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Köln, Cologne
  - BAG Freiberg-Richter, Jacobasch, Illmer, Wolf, Dresden
  - Uniklinikum "Carl Gustav Carus";Med. Klinik 1, Dresden
  - Universitätsklinikum Essen, Essen
  - Klinik Esslingen, Esslingen am Neckar
  - Klinikum Frankfurt/Oder, Frankfurt (Oder)
  - Uniklinikum Freiburg, Freiburg im Breisgau
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Stiftung Kathol. Krankenhaus Marienhospital Herne Klinik Mitte, Herne
  - Praxisklinik für Hämatologie und Onkologie Koblenz, Koblenz
  - Kliniken Maria Hilf GmbH Innere Medizin I, Mönchengladbach
  - Klinikum Schwäbisch Gmünd, Mutlangen
  - München Klinik Schwabing, München
  - Klinikum rechts der Isar der Technischen Universität München, München
  - Klinikum der Universität München, Campus Großhadern, München
  - Brüderkrankenhaus St. Josef Paderborn, Paderborn
  - Krankenhaus Barmherzige Bruder Regensburg, Regensburg
  - Marienhospital, Stuttgart
  - Robert-Bosch-Krankenhaus, Stuttgart
  - Universitatsklinikum Tubingen, Tübingen
  - Universtitätsklinikum Ulm, Ulm
- Italy (6):
  - Arcispedale S. Anna, Ferrara, Emilia-Romagna
  - Uni Cattolica, Rome, Lazio
  - AOU Città della Salute e della Scienza di Torino - Presidio Le Molinette, Torino, Lazio
  - Ospedale San Raffaele, Milan, Lombardy
  - Az. Osp. S. Maria, Terni, Umbria
  - Ospedale dell' Angelo, Venezia Mestre, Veneto
- Hospital General de Culiacan, Culiacán, Sinaloa, Mexico
- New Zealand (4):
  - Canterbury Health Laboratories, Christchurch
  - Dunedin Hospital, Dunedin
  - Midcentral District Health Board, Palmerston North
  - Wellington Hospital, Wellington
- Poland (4):
  - Samodzielny Public Zaklad, Chorzów
  - Wojewódzki Szpital Specjalistyczny im. Miko?aja Kopernika, Lodz
  - Wojewodzki Szpital Specjalistyczny im. J. Korczaka, Słupsk
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 we Wroc?awiu, Wroclaw
- Romania (3):
  - Fundeni Clinical Inst., Bucharest
  - Institutul Regional de Oncologie Iasi, Iași
  - Spitalul Clinic Judetean de Urgenta Targu-Mures, Târgu Mureş
- Russia (5):
  - SBEI of HPE ?Bashkir State Medical University? of MoH RF, Ufa, Bashkortostan Republic
  - Regional Clinical Hospital N.A. Semashko, Nizhny Novgorod, Niznij Novgorod
  - Republican Clinical Oncologic Dispensary of Republic Of Tatarstan, Kazan', Tatarstan Republic
  - Penza Regional Oncology Dispensary, Penza
  - Clinical MSCh No1, Perm
- Spain (14):
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Tenerife
  - Hospital del Mar, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clínic i Provincial, Barcelona
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Univ. 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocio, Seville
  - Complejo Hospitalario de Toledo- H. Virgen de la Salud, Toledo
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Arnau de Vilanova (Valencia) Servicio de Hematologia, Valencia
- Switzerland (3):
  - Inselspital Bern, Bern
  - Luzerner Kantonsspital, Hämatologie, Lucerne
  - Universitätsspital Zürich Medizin Hämatologie, Zurich
- United Kingdom (5):
  - Birmingham Heartlands Hospital, Birmingham
  - Boston Pilgrim Hospital, Boston,Lincolnshire
  - Western General Hospital, Edinburgh
  - Lincoln County Hospital, Lincoln
  - University Hospital Southampton NHS Foundation Trust, Southhampton

REFERENCES:
- [Derived] Munir T, Martinez-Calle N, Xu S, Yang K, Ge X, Ali AK, Mohseninejad L, Dobi B, Rakonczai P, Ma H, Williams R, Aldairy W, Lamanna N. Indirect Comparisons of the Efficacy and Safety of Zanubrutinib versus Venetoclax plus Obinutuzumab in Treatment-Naive Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma. Oncol Ther. 2025 Dec;13(4):1055-1070. doi: 10.1007/s40487-025-00380-0. Epub 2025 Sep 13. PMID 40944848
- [Derived] Al-Sawaf O, Robrecht S, Zhang C, Olivieri S, Chang YM, Fink AM, Tausch E, Schneider C, Ritgen M, Kreuzer KA, Sivchev L, Niemann CU, Schwarer A, Loscertales J, Weinkove R, Strumberg D, Kilfoyle A, Manzoor BS, Jawaid D, Emechebe N, Devine J, Boyer M, Runkel ED, Eichhorst B, Stilgenbauer S, Jiang Y, Hallek M, Fischer K. Venetoclax-obinutuzumab for previously untreated chronic lymphocytic leukemia: 6-year results of the randomized phase 3 CLL14 study. Blood. 2024 Oct 31;144(18):1924-1935. doi: 10.1182/blood.2024024631. PMID 39082668
- [Derived] Langerbeins P, Giza A, Robrecht S, Cramer P, von Tresckow J, Al-Sawaf O, Fink AM, Furstenau M, Kutsch N, Simon F, Goede V, Hoechstetter M, Niemann CU, da Cunha-Bang C, Kater A, Dubois J, Gregor M, Staber PB, Tausch E, Schneider C, Stilgenbauer S, Eichhorst B, Fischer K, Hallek M. Reassessing the chronic lymphocytic leukemia International Prognostic Index in the era of targeted therapies. Blood. 2024 Jun 20;143(25):2588-2598. doi: 10.1182/blood.2023022564. PMID 38620092
- [Derived] Al-Sawaf O, Zhang C, Jin HY, Robrecht S, Choi Y, Balasubramanian S, Kotak A, Chang YM, Fink AM, Tausch E, Schneider C, Ritgen M, Kreuzer KA, Chyla B, Paulson JN, Pallasch CP, Frenzel LP, Peifer M, Eichhorst B, Stilgenbauer S, Jiang Y, Hallek M, Fischer K. Transcriptomic profiles and 5-year results from the randomized CLL14 study of venetoclax plus obinutuzumab versus chlorambucil plus obinutuzumab in chronic lymphocytic leukemia. Nat Commun. 2023 Apr 18;14(1):2147. doi: 10.1038/s41467-023-37648-w. PMID 37072421
- [Derived] Badawi M, Chen X, Marroum P, Suleiman AA, Mensing S, Koenigsdorfer A, Schiele JT, Palenski T, Samineni D, Hoffman D, Menon R, Salem AH. Bioavailability Evaluation of Venetoclax Lower-Strength Tablets and Oral Powder Formulations to Establish Interchangeability with the 100 mg Tablet. Clin Drug Investig. 2022 Aug;42(8):657-668. doi: 10.1007/s40261-022-01172-4. Epub 2022 Jul 13. PMID 35829925
- [Derived] Samineni D, Gibiansky L, Wang B, Vadhavkar S, Rajwanshi R, Tandon M, Sinha A, Al-Sawaf O, Fischer K, Hallek M, Salem AH, Li C, Miles D. Pharmacokinetics and Exposure-Response Analysis of Venetoclax + Obinutuzumab in Chronic Lymphocytic Leukemia: Phase 1b Study and Phase 3 CLL14 Trial. Adv Ther. 2022 Aug;39(8):3635-3653. doi: 10.1007/s12325-022-02170-w. Epub 2022 Jun 16. PMID 35708885
- [Derived] Al-Sawaf O, Zhang C, Lu T, Liao MZ, Panchal A, Robrecht S, Ching T, Tandon M, Fink AM, Tausch E, Schneider C, Ritgen M, Bottcher S, Kreuzer KA, Chyla B, Miles D, Wendtner CM, Eichhorst B, Stilgenbauer S, Jiang Y, Hallek M, Fischer K. Minimal Residual Disease Dynamics after Venetoclax-Obinutuzumab Treatment: Extended Off-Treatment Follow-up From the Randomized CLL14 Study. J Clin Oncol. 2021 Dec 20;39(36):4049-4060. doi: 10.1200/JCO.21.01181. Epub 2021 Oct 28. PMID 34709929
- [Derived] Al-Sawaf O, Zhang C, Tandon M, Sinha A, Fink AM, Robrecht S, Samoylova O, Liberati AM, Pinilla-Ibarz J, Opat S, Sivcheva L, Le Du K, Fogliatto LM, Niemann CU, Weinkove R, Robinson S, Kipps TJ, Tausch E, Schary W, Ritgen M, Wendtner CM, Kreuzer KA, Eichhorst B, Stilgenbauer S, Hallek M, Fischer K. Venetoclax plus obinutuzumab versus chlorambucil plus obinutuzumab for previously untreated chronic lymphocytic leukaemia (CLL14): follow-up results from a multicentre, open-label, randomised, phase 3 trial. Lancet Oncol. 2020 Sep;21(9):1188-1200. doi: 10.1016/S1470-2045(20)30443-5. PMID 32888452
- [Derived] Fischer K, Al-Sawaf O, Bahlo J, Fink AM, Tandon M, Dixon M, Robrecht S, Warburton S, Humphrey K, Samoylova O, Liberati AM, Pinilla-Ibarz J, Opat S, Sivcheva L, Le Du K, Fogliatto LM, Niemann CU, Weinkove R, Robinson S, Kipps TJ, Boettcher S, Tausch E, Humerickhouse R, Eichhorst B, Wendtner CM, Langerak AW, Kreuzer KA, Ritgen M, Goede V, Stilgenbauer S, Mobasher M, Hallek M. Venetoclax and Obinutuzumab in Patients with CLL and Coexisting Conditions. N Engl J Med. 2019 Jun 6;380(23):2225-2236. doi: 10.1056/NEJMoa1815281. Epub 2019 Jun 4. PMID 31166681

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Obinutuzumab + Chlorambucil | Obinutuzumab + Venetoclax | Safety Run-in Obinutuzumab + Venetoclax
Started | 216 | 216 | 13
Treated | 214 | 212 | 13
Completed | 0 | 0 | 0
Not Completed | 216 | 216 | 13
Not completed — Death | 17 | 20 | 2
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Withdrawal by Subject | 8 | 10 | 0
Not completed — On-going in Study | 190 | 186 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Obinutuzumab + Chlorambucil | Obinutuzumab + Venetoclax | Safety Run-in Obinutuzumab + Venetoclax | Total
Number analyzed (Participants) | 216 | 216 | 13 | 445
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.1 (8.0) | 71.1 (8.2) | 75.4 (7.8) | 71.1 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 70 | 5 | 148
  Male | 143 | 146 | 8 | 297
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 22 | 1 | 43
  Not Hispanic or Latino | 172 | 165 | 12 | 349
  Not Stated | 19 | 22 | 0 | 41
  Unknown | 5 | 7 | 0 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Black or African American | 3 | 1 | 0 | 4
  Native Hawaiian or other Pacific Islande | 0 | 3 | 0 | 3
  Unknown | 18 | 20 | 0 | 38
  White | 194 | 192 | 13 | 399

OUTCOME MEASURES:

1. Secondary Outcome: Progression Free Survival (PFS) Based on Institutional Review Committee (IRC)-Assessments According to International Workshop on Chronic Lymphocytic Leukemia (IWCLL) Criteria
Description: PFS was determined according to IWCLL 2008 criteria and defined as the time from randomization to the first occurrence of progressive disease (PD) or death from any cause. Disease progression was characterized by at least one of the following: 1) >/= 50% increase in the absolute number of circulating lymphocytes to at least 5*10^9/L, 2) Appearance of new palpable lymph nodes (> 15 mm in longest diameter) or any new extra-nodal lesion; 3) >/= 50% increase in the longest diameter of any previous site of lymphadenopathy; 4) >/= 50% increase in the enlargement of the liver and/or spleen; 5) Transformation to a more aggressive histology.
Time Frame: Baseline until disease progression or death up to approximately 3.75 years
Population: Intent-to-Treat (ITT) population was defined as all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Obinutuzumab + Chlorambucil: Participants received obinutuzumab for 6 cycles and chlorambucil for 12 cycles. Cycles comprised 28 days.
- Obinutuzumab + Venetoclax: Participants received obinutuzumab for 6 cycles and venetoclax for 12 cycles. Cycles comprised 28 days.
Arm/Group | Obinutuzumab + Chlorambucil | Obinutuzumab + Venetoclax
Number analyzed (Participants) | 216 | 216
months | NA [31.1 to NA] — Insufficient number of participants with events. | NA [NA to NA] — Insufficient number of participants with events.
Statistical Analysis 1: Comparison: Obinutuzumab + Chlorambucil vs Obinutuzumab + Venetoclax; Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.33, 95% CI 2-sided [0.22 to 0.51] — Hazard ratios were estimated by Cox regression model. Stratification factors: Binet and Geographic region

2. Primary Outcome: Progression Free Survival (PFS) Based on Investigator Assessment According to IWCLL Criteria
Description: PFS was determined according to IWCLL 2008 criteria and defined as the time from randomization to the first occurrence of PD or death from any cause. Disease progression was characterized by at least one of the following: 1) >/= 50% increase in the absolute number of circulating lymphocytes to at least 5*10^9/L, 2) Appearance of new palpable lymph nodes (> 15 mm in longest diameter) or any new extra-nodal lesion; 3) >/= 50% increase in the longest diameter of any previous site of lymphadenopathy; 4) >/= 50% increase in the enlargement of the liver and/or spleen; 5) Transformation to a more aggressive histology.
Time Frame: Baseline until disease progression or death up to approximately 3.75 years
Population: ITT population was defined as all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Obinutuzumab + Chlorambucil | Obinutuzumab + Venetoclax
Number analyzed (Participants) | 216 | 216
months | NA [31.1 to NA] — Insufficient number of participants with events. | NA [NA to NA] — Insufficient number of participants with events.
Statistical Analysis 1: Comparison: Obinutuzumab + Chlorambucil vs Obinutuzumab + Venetoclax; Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.35, 95% CI 2-sided [0.23 to 0.53] — Hazard Ratios were estimated by Cox regression model. Stratification factors: Binet and Geographic region

3. Secondary Outcome: Percentage of Participants With an Overall Response (OR) at Completion of Treatment, as Determined by the Investigator According to IWCLL Criteria
Description: OR was defined as complete response (CR), CR with incomplete bone marrow recovery (CRi), or partial response (PR) according to IWCLL 2008 criteria. CR requires all of the following: peripheral blood lymphocytes below 4x10^9/L, absence of lymphadenopathy by physical examination and computed tomography (CT) scan, no hepatomegaly or splenomegaly, absence of disease or constitutional symptoms, blood counts of neutrophils >1.5*10^9/L, platelets >100*10^9/L and hemoglobin >110 g/L, bone marrow at least normocellular for age without clonal infiltrate (except for Cri). PR: two of the following features for at least 2 months: >/= 50% decrease in peripheral blood lymphocyte count from the pretreatment value, >/=50% reduction in lymphadenopathy, >/=50% reduction of liver and/or spleen enlargement, and at least one of the following blood counts: neutrophils >1.5*10^9/L, platelets >100*10^9/L and hemoglobin >110 g/L.
Time Frame: At the completion of treatment assessment 3 months after treatment completion (at approximately 15 months)
Population: ITT population was defined as all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Obinutuzumab + Chlorambucil | Obinutuzumab + Venetoclax
Number analyzed (Participants) | 216 | 216
percentage of participants | 71.3 [64.77 to 77.23] | 84.7 [79.22 to 89.24]
Statistical Analysis 1: Comparison: Obinutuzumab + Chlorambucil vs Obinutuzumab + Venetoclax; Test type: Superiority; p = 0.0007, Cochran-Mantel-Haenszel — P-value was assessed using Cochran-Mantel-Haenszel (CMH) test stratified by the IvRS randomization stratification factors; Difference in Response Rates = 13.43, 95% CI 2-sided [5.47 to 21.38] — 95% Confidence Interval (CI) for difference in rates were constructed using Anderson-Hauck method

4. Secondary Outcome: Percentage of Participants With a Complete Response Rate (CRR) at the Completion of Treatment Assessment as Determined by the Investigator According to IWCLL Criteria
Description: CRR was defined as the rate of a clinical response of CR or CRi according to IWCLL 2008 criteria. CR requires all of the following: peripheral blood lymphocytes below 4x10^9/L, absence of lymphadenopathy by physical examination and CT scan, no hepatomegaly or splenomegaly, absence of disease or constitutional symptoms, blood counts of neutrophils >1.5*10^9/L, platelets >100*10^9/L and hemoglobin >110 g/L, bone marrow at least normocellular for age without clonal infiltrate (except for Cri).
Time Frame: At the completion of treatment assessment 3 months after treatment completion (at approximately 15 months)
Population: ITT population was defined as all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Obinutuzumab + Chlorambucil | Obinutuzumab + Venetoclax
Number analyzed (Participants) | 216 | 216
percentage of participants | 23.1 [17.70 to 29.35] | 49.5 [42.68 to 56.40]
Statistical Analysis 1: Comparison: Obinutuzumab + Chlorambucil vs Obinutuzumab + Venetoclax; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was assessed using CMH test stratified by the IvRS randomization stratification factors; Difference in Response Rates = 26.39, 95% CI 2-sided [17.41 to 35.36] — 95% CI for difference in rates were constructed using Anderson-Hauck method

5. Secondary Outcome: Percentage of Participants With Minimal Residual Disease (MRD) Negativity in Peripheral Blood as Measured by Allele-Specific Oligonucleotide Polymerase Chain Reaction (ASO-PCR) at Completion of Treatment
Description: MRD negativity was defined as having < 1 CLL cell per 10,000 leucocytes in peripheral blood.
Time Frame: At the completion of treatment assessment 3 months after treatment completion (at approximately 15 months)
Population: ITT population was defined as all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Obinutuzumab + Chlorambucil | Obinutuzumab + Venetoclax
Number analyzed (Participants) | 216 | 216
percentage of participants | 35.2 [28.83 to 41.95] | 75.5 [69.17 to 81.05]
Statistical Analysis 1: Comparison: Obinutuzumab + Chlorambucil vs Obinutuzumab + Venetoclax; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in MRD Negative Rates = 40.28, 95% CI 2-sided [31.45 to 49.10] — 95% CI for difference in rates were constructed using Anderson-Hauck method

6. Secondary Outcome: Percentage of Participants With MRD Negativity in Bone Marrow as Measured by ASO-PCR at Completion of Treatment
Description: MRD negativity was defined as having < 1 CLL cell per 10,000 leucocytes in bone marrow.
Time Frame: At the completion of treatment assessment 3 months after treatment completion (at approximately 15 months)
Population: ITT population was defined as all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Obinutuzumab + Chlorambucil | Obinutuzumab + Venetoclax
Number analyzed (Participants) | 216 | 216
percentage of participants | 17.1 [12.36 to 22.83] | 56.9 [50.05 to 63.64]
Statistical Analysis 1: Comparison: Obinutuzumab + Chlorambucil vs Obinutuzumab + Venetoclax; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in MRD Negative Rates = 39.81, 95% CI 2-sided [31.27 to 48.36] — 95% CI for difference in rates were constructed using Anderson-Hauck method

7. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time between the date of randomization and the date of death due to any cause.
Time Frame: Baseline until death, up to approximately 10.75 years
Reporting Status: Not Posted, anticipated posting 2026-08

8. Secondary Outcome: Percentage of Participants With MRD Negativity in Peripheral Blood as Measured by ASO-PCR at Completion of Combination Treatment Assessment
Description: MRD negativity was defined as having < 1 CLL cell per 10,000 leucocytes in peripheral blood.
Time Frame: Day 1 Cycle 9 or 3 months after last IV infusion, approximately 9 months
Population: ITT population was defined as all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Obinutuzumab + Chlorambucil | Obinutuzumab + Venetoclax
Number analyzed (Participants) | 216 | 216
percentage of participants | 38.4 [31.91 to 45.27] | 71.3 [64.77 to 77.23]
Statistical Analysis 1: Comparison: Obinutuzumab + Chlorambucil vs Obinutuzumab + Venetoclax; Test type: Superiority; p < 0.0001, Chi-squared; Difference in MRD Negative Rates = 32.87, 95% CI 2-sided [23.76 to 41.98] — 95% CI for difference in rates were constructed using Anderson-Hauck method

9. Secondary Outcome: Percentage of Participants With MRD Negativity in Bone Marrow as Measured by ASO-PCR at Completion of Combination Treatment Assessment
Description: MRD negativity was defined as having < 1 CLL cell per 10,000 leucocytes in bone marrow.
Time Frame: Day 1 Cycle 9 or 3 months after last IV infusion at approximately 9 months
Population: ITT population was defined as all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Obinutuzumab + Chlorambucil | Obinutuzumab + Venetoclax
Number analyzed (Participants) | 216 | 216
percentage of participants | 13.0 [8.79 to 18.19] | 51.4 [44.51 to 58.23]
Statistical Analysis 1: Comparison: Obinutuzumab + Chlorambucil vs Obinutuzumab + Venetoclax; Test type: Superiority; p < 0.0001, Chi-squared; Difference in MRD Negative Rates = 38.43, 95% CI 2-sided [30.15 to 46.71] — 95% CI for difference in rates were constructed using Anderson-Hauck method

10. Secondary Outcome: Percentage of Participants With OR at Completion of Combination Treatment Response Assessment
Description: OR was defined as CR, CRi or PR according to IWCLL 2008 criteria. CR required all of the following: peripheral blood lymphocytes below 4x10^9/L, absence of lymphadenopathy by physical examination, no hepatomegaly or splenomegaly, absence of disease or constitutional symptoms, blood counts of neutrophils >1.5*10^9/L, platelets >100*10^9/L and hemoglobin >110 g/L. PR: two of the following features for at least 2 months: >/= 50% decrease in peripheral blood lymphocyte count from the pretreatment value, >/=50% reduction in lymphadenopathy, >/=50% reduction of liver and/or spleen enlargement, and at least one of the following blood counts: neutrophils >1.5*10^9/L, platelets >100*10^9/L and hemoglobin >110 g/L.
Time Frame: Day 1 Cycle 7 or 28 days after last IV infusion, approximately 6 months
Population: ITT population was defined as all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Obinutuzumab + Chlorambucil | Obinutuzumab + Venetoclax
Number analyzed (Participants) | 216 | 216
percentage of participants | 86.6 [81.29 to 90.82] | 88.4 [83.39 to 92.37]
Statistical Analysis 1: Comparison: Obinutuzumab + Chlorambucil vs Obinutuzumab + Venetoclax; Test type: Superiority; p = 0.5612, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Difference in Response Rates = 1.85, 95% CI 2-sided [-4.63 to 8.33] — 95% Confidence Interval (CI) for difference in rates were constructed using Anderson-Hauck method

11. Secondary Outcome: Duration of Objective Response (DOR)
Description: PD was defined as lymphadenopathy, >=50% increase in liver or spleen size, >=50% increase in lymphocyte count, transformation to a more aggressive histology or occurrence of cytopenia.
Time Frame: Time from the first occurrence of a documented objective response to the time of PD as determined by the investigator or death from any cause, up to approximately 10.75 years
Reporting Status: Not Posted, anticipated posting 2026-08

12. Secondary Outcome: Percentage of Participants By Best Response Achieved (CR, CRi, PR, Stable Disease (SD), or PD)
Description: CR: peripheral blood lymphocytes below 4x10^9/L, absence of lymphadenopathy by physical examination and CT scan, no hepatomegaly or splenomegaly, absence of disease or constitutional symptoms, blood counts of neutrophils >1.5*10^9/L, platelets >100*10^9/L and hemoglobin >110 g/L, bone marrow at least normocellular for age without clonal infiltrate (except for Cri). PR: any two for at least 2 months: >/= 50% decrease in peripheral blood lymphocyte count from the pretreatment value, >/=50% reduction in lymphadenopathy, >/=50% reduction of liver and/or spleen enlargement, and at least one of the following blood counts: neutrophils >1.5*10^9/L, platelets >100*10^9/L and hemoglobin >110 g/L. PD: lymphadenopathy, >=50% increase in liver or spleen size, >=50% increase in lymphocyte count, transformation to a more aggressive histology or occurrence of cytopenia. SD: a non-response and used to characterize participants who did not achieve a CR or a PR, and who have not exhibited PD.
Time Frame: Baseline up to the completion of treatment assessment 3 months after treatment completion (up to approximately 15 months)
Population: ITT population was defined as all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Obinutuzumab + Chlorambucil | Obinutuzumab + Venetoclax
Number analyzed (Participants) | 216 | 216
percentage of participants
  CR | 56.0 | 70.4
  CRi | 5.6 | 7.9
  PR | 29.2 | 13.4
  SD | 1.9 | 0.5
  PD | 0.5 | 0.5
Statistical Analysis 1: Comparison: Obinutuzumab + Chlorambucil vs Obinutuzumab + Venetoclax; Test type: Superiority; p = 0.7169, Cochran-Mantel-Haenszel; P-value was assessed using CMH test stratified by the IvRS randomization stratification factors; Difference in Response Rates = 0.93, 95% CI 2-sided [-4.66 to 6.51] — 95% CI for difference in rates were constructed using Anderson-Hauck method

13. Secondary Outcome: Event-Free Survival
Time Frame: Time between date of randomization and the date of disease progression/relapse on the basis of investigator-assessment, death, or start of a new anti-leukemic therapy, up to 10.75 years
Reporting Status: Not Posted, anticipated posting 2026-08

14. Secondary Outcome: Time to Next Anti-Leukemic Treatment
Time Frame: Time between the date of randomization and the date of first intake of new anti-leukemic therapy, up to 10.75 years
Reporting Status: Not Posted, anticipated posting 2026-08

15. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as AEs.
Time Frame: Up to approximately 10.75 years
Reporting Status: Not Posted, anticipated posting 2026-08

16. Secondary Outcome: Percentage of Participants With CD19 + /CD5+ B Cells or CD14+ Monocytes
Time Frame: Baseline up to approximately 10.75 years
Reporting Status: Not Posted, anticipated posting 2026-08

17. Secondary Outcome: Percentage of Participants With Human-Anti-Human Antibodies
Time Frame: Baseline up to approximately 10.75 years
Reporting Status: Not Posted, anticipated posting 2026-08

18. Secondary Outcome: Percentage of Participants Recorded as Premature Study Withdrawals
Time Frame: Up to approximately 10.75 years
Reporting Status: Not Posted, anticipated posting 2026-08

19. Secondary Outcome: Plasma Concentrations of Venetoclax
Time Frame: Pre-venetoclax dose (0 hour) and 4 hours post- venetoclax dose on Day 1 Cycle 4
Population: Analysis population consisted of subjects from whom one or more plasma samples were collected and who had received at least one 400 mg dose of venetoclax. Pre-dose and post-dose data may not come from the same participants. Total number analyzed is therefore higher than the number analyzed for each time point.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Obinutuzumab + Venetoclax
Number analyzed (Participants) | 184
μg/mL
  Pre-Dose: number analyzed (Participants) | 129
  Pre-Dose | 0.578 (0.533)
  4 hours Post-Dose: number analyzed (Participants) | 142
  4 hours Post-Dose | 1.21 (0.765)

20. Secondary Outcome: Serum Concentrations of Obinutuzumab
Time Frame: Pre-obinutuzumab infusion (0 hour) and end of obinutuzumab infusion on Day 1 Cycle 4
Population: Analysis population consisted of subjects from whom one or more serum samples were collected and who had received at least one dose of obinutuzumab and one dose of 400 mg venetoclax. Pre-dose and post-dose data may not come from the same participants. Total number analyzed is therefore higher than the number analyzed for each time point.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Obinutuzumab + Venetoclax
Number analyzed (Participants) | 184
μg/mL
  Pre-Dose: number analyzed (Participants) | 133
  Pre-Dose | 258 (140)
  4 hours Post-Dose: number analyzed (Participants) | 133
  4 hours Post-Dose | 568 (187)

21. Secondary Outcome: Change From Baseline in M.D. Anderson Symptom Inventory-CLL (MDASI-CLL) Score
Description: The MDASI-CLL is a questionnaire of 25 items related to CLL specific symptoms that a participant may have experienced in the past 24 hours. Participants were asked to rate the severity of 13 symptoms called mean core symptom severity (i.e., pain, fatigue, nausea, disturbed sleep, distressed, shortness of breath, remembering things, lack of appetite, drowsy, dry mouth, sadness, vomiting, and numbness or tingling), 6 disease-specific symptoms called mean module symptom severity (night sweats, fevers and chills, lymph node swelling, diarrhea, easy bruising or bleeding, and constipation) and 6 mean interference on life questions (i.e., general activity, walking, work, mood, relations with other people, and enjoyment of life) on a scale from 0 to 10 with 0 indicating that the symptom is "not present" or "did not interfere" with the participant's activities and 10 indicating "as bad as you can imagine" or "interfered completely". Scores were averaged (range 0 to 10) for each of three parts.
Time Frame: Baseline up to approximately 10.75 years
Reporting Status: Not Posted, anticipated posting 2026-08

22. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQC30)
Description: The EORTC QLQ-C30 is a validated and reliable self-report measure consisting of 30 questions incorporated into five functional scales (physical, role, cognitive, emotional, and social scales), three symptom scales (fatigue, pain, nausea, and vomiting scales), and a global health status/global quality-of-life scale. The remaining single items (dyspnea, appetite loss, sleep disturbance, constipation, and diarrhea) assess the additional symptoms experienced by patients with cancer and the perceived financial burden of treatment. The 28 function and symptom items were scored on a 4-point scale that ranged from "not at all" to "very much," and the 2 global health status/global quality-of-life items were scored on a 7-point scale that ranged from "very poor" to "excellent." Raw average scale scores were linearly transformed to range 0-100 with higher scores indicating higher response levels (i.e., higher functioning, higher symptom severity).
Time Frame: Baseline up to approximately 10.75 years
Reporting Status: Not Posted, anticipated posting 2026-08

23. Secondary Outcome: Change From Baseline in EuroQol 5 Dimension Questionnaire (EQ-5D-3L)
Description: The EQ-5D-3L questionnaire is a generic, preference based health utility measure that assesses 5 health states (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) and is used to build a composite of the patient's health status. The EQ-5D-3L was employed in this study to calculate health utilities for economic modeling, which ranged 0-1. The EQ-5D-3L also contained a visual analog scale (VAS) to assess the participant's overall health, which ranged from 0-100 with a higher score indicating a worse health status.
Time Frame: Baseline up to approximately 10.75 years
Reporting Status: Not Posted, anticipated posting 2026-08

ADVERSE EVENTS:
Time Frame: All AEs from first dose until 28 days after the last dose up to 1 year. Grade 3-4 AEs: for 6 months after last dose (up to 1.5 years). Major infections (Grade 3-4): for 2 years after the last dose (up to 3 years) irrespective of causality unless disease progressed and participant received leukemic treatment. Before disease progression, SAEs were reported during follow-up (up to 3.75 years). After disease progression, only related SAEs and second primary malignancies were reported.
Description: All-cause mortality was based on the ITT population defined as all randomized participants. Reporting of serious and non-serious adverse events was based on the safety population defined as all participants who received at least one dose of any study medication (i.e., obinutuzumab, venetoclax, or chlorambucil).
Arm/Group | Obinutuzumab + Chlorambucil | Obinutuzumab + Venetoclax | Safety Run-in Obinutuzumab + Venetoclax
All-Cause Mortality (participants affected / at risk) | 17/216 | 20/216 | 2/13
Serious Adverse Events (participants affected / at risk) | 90/214 | 104/212 | 10/13
Other Adverse Events (participants affected / at risk) | 205/214 | 193/212 | 12/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Obinutuzumab + Chlorambucil (N=214) | Obinutuzumab + Venetoclax (N=212) | Safety Run-in Obinutuzumab + Venetoclax (N=13)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (3) | 0 (0)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Coombs negative haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 8 (10) | 11 (12) | 3 (3)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (5) | 2 (2) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 2 (3) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 3 (3) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 3 (4) | 1 (1) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Gilbert's syndrome (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0)
Amaurosis fugax (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eye inflammation (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (2) | 2 (2) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Adverse drug reaction (General disorders) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1)
Device related thrombosis (General disorders) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 7 (8) | 8 (8) | 2 (2)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Cholecystitis infective (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Eczema infected (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hepatitis E (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 2 (2) | 2 (4) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Listeriosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Muscle abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Neutropenic infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ophthalmic herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 9 (11) | 10 (10) | 1 (1)
Pneumonia fungal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia haemophilus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 6 (7) | 1 (2)
Septic shock (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Sinusitis aspergillus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (2) | 2 (2) | 0 (0)
Varicella zoster virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Wound infection fungal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Chillblains (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 13 (13) | 9 (9) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Vasoplegia syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound evisceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (3) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Prothrombin time prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Penile cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Sarcoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Skin squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2) | 0 (0)
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (2) | 1 (1)
Vertebrobasilar insufficiency (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (10) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Aortic valve replacement (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Medical device removal (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Obinutuzumab + Chlorambucil (N=214) | Obinutuzumab + Venetoclax (N=212) | Safety Run-in Obinutuzumab + Venetoclax (N=13)
Anaemia (Blood and lymphatic system disorders) | 39 (55) | 33 (53) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 13 (19) | 12 (23) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 122 (294) | 121 (370) | 8 (12)
Thrombocytopenia (Blood and lymphatic system disorders) | 49 (76) | 49 (86) | 2 (5)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 5 (5) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Excessive cerumen production (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 10 (11) | 11 (15) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4) | 7 (7) | 1 (1)
Constipation (Gastrointestinal disorders) | 19 (23) | 28 (32) | 5 (6)
Diarrhoea (Gastrointestinal disorders) | 32 (42) | 59 (99) | 5 (8)
Dry mouth (Gastrointestinal disorders) | 4 (4) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 7 (7) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 46 (62) | 40 (61) | 4 (7)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (2)
Vomiting (Gastrointestinal disorders) | 18 (22) | 21 (27) | 3 (3)
Adverse drug reaction (General disorders) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 17 (20) | 14 (20) | 0 (0)
Chills (General disorders) | 10 (13) | 12 (14) | 1 (1)
Extravasation (General disorders) | 2 (2) | 0 (0) | 1 (1)
Fatigue (General disorders) | 29 (36) | 32 (40) | 3 (6)
Influenza like illness (General disorders) | 3 (3) | 4 (4) | 1 (1)
Oedema (General disorders) | 7 (7) | 3 (3) | 1 (1)
Oedema peripheral (General disorders) | 16 (18) | 17 (20) | 1 (2)
Pyrexia (General disorders) | 26 (28) | 40 (53) | 3 (4)
Sensation of foreign body (General disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 5 (6) | 11 (14) | 1 (2)
Cystitis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Eye infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (3)
Herpes zoster (Infections and infestations) | 6 (7) | 9 (9) | 1 (1)
Influenza (Infections and infestations) | 4 (4) | 3 (3) | 1 (1)
Localised infection (Infections and infestations) | 3 (3) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 14 (16) | 16 (16) | 0 (0)
Oral herpes (Infections and infestations) | 4 (5) | 5 (7) | 1 (4)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 6 (9) | 1 (1)
Respiratory tract infection (Infections and infestations) | 6 (7) | 10 (14) | 1 (3)
Rhinitis (Infections and infestations) | 5 (6) | 2 (3) | 1 (1)
Sinusitis (Infections and infestations) | 6 (6) | 8 (8) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 15 (17) | 16 (19) | 2 (4)
Urinary tract infection (Infections and infestations) | 9 (10) | 10 (13) | 1 (1)
Viral skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 8 (11) | 5 (7) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 103 (131) | 89 (122) | 9 (10)
Limb injury (Injury, poisoning and procedural complications) | 4 (4) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1)
Alanine aminotransferase increased (Investigations) | 13 (15) | 11 (15) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 17 (20) | 12 (14) | 0 (0)
Blood albumin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 6 (6) | 7 (9) | 1 (2)
Blood glucose increased (Investigations) | 1 (1) | 1 (1) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 2 (2) | 2 (2) | 2 (2)
Blood magnesium decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood phosphorus increased (Investigations) | 1 (1) | 2 (4) | 1 (1)
C-reactive protein increased (Investigations) | 2 (2) | 4 (4) | 1 (1)
Neutrophil count decreased (Investigations) | 11 (32) | 10 (27) | 0 (0)
Procalcitonin increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Protein total decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 2 (2) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 5 (5) | 5 (5) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 6 (8) | 10 (10) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (2) | 3 (4) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 7 (7) | 14 (16) | 2 (4)
Hyperkalaemia (Metabolism and nutrition disorders) | 5 (6) | 4 (13) | 5 (7)
Hyperphosphataemia (Metabolism and nutrition disorders) | 3 (3) | 4 (5) | 1 (1)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 (23) | 16 (19) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 20 (21) | 21 (24) | 2 (2)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 11 (11) | 10 (11) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (4) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 7 (8) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 (14) | 10 (11) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (6) | 6 (6) | 1 (1)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 17 (20) | 16 (18) | 4 (5)
Headache (Nervous system disorders) | 21 (24) | 23 (29) | 3 (3)
Paraesthesia (Nervous system disorders) | 1 (1) | 4 (4) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1) | 2 (3)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 4 (4) | 5 (5) | 2 (2)
Tremor (Nervous system disorders) | 3 (4) | 6 (6) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 8 (8) | 1 (1)
Dysuria (Renal and urinary disorders) | 2 (2) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (3)
Renal impairment (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 24 (27) | 33 (37) | 6 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 11 (12) | 1 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (3) | 1 (1)
Pharyngeal paraesthesia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (6) | 1 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (7) | 4 (4) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (9) | 18 (20) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 12 (13) | 12 (12) | 2 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 3 (3) | 2 (2) | 2 (2)
Hypertension (Vascular disorders) | 11 (12) | 12 (17) | 0 (0)
Hypotension (Vascular disorders) | 8 (10) | 11 (15) | 2 (2)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-02-12): https://cdn.clinicaltrials.gov/large-docs/42/NCT02242942/Prot_001.pdf
  • Statistical Analysis Plan (2018-11-08): https://cdn.clinicaltrials.gov/large-docs/42/NCT02242942/SAP_000.pdf